CLINICAL TRIAL: NCT01644539
Title: Functional MRI of Satiety, the Interaction Between Gastric and Oral Stimulation and Related Hormones in Healthy Men
Brief Title: Brain Activity and Hormonal Changes During Food Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Paul A.M. Smeets, Principal investigator, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL 35991.041.11
Record Dates: First submitted 2012-07-12; First posted 2012-07-19 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Appetite Regulation
Keywords: Satiation; Brain activation; Gut peptides
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Other): Subjects participated in a 35 min fmri scan. Intervention: intra-gastric infusion of 500 ml non caloric load consisting of water and thickening agent (guar gum), over 5 min.
  While scanning:
  -5 - 0 min : baseline scan 0 - 5 min: intra-gastric infusion (naso-gastric tube) of 500 ml non caloric load consisting of water and thickening agent (guar gum) in a time frame of 5 minutes while being scanned (fmri) 5 - 30 min: fmri scan continues while subject lays still
  At t = 0, 2.5, 5, 10, 15 and 30 blood will be drawn and appetite ratings will be given.
  Interventions: Dietary Supplement: Water with guar gum - Non Caloric
- Oral ingestion (Other): Subjects participated in a 35 min fmri scan. Intervention: Oral ingestion (through a tube, while drinking and swallowing on command) of 500 ml caloric load consisting of Nutricia Chocolate Milk, over 5 min.
  Time frame while scanning:
  -5 - 0 min : baseline fmri scan 0 - 5 min: oral ingestion (through a tube, while drinking and swallowing on command) of 500 ml caloric load consisting of Nutricia Chocolate Milk in a time frame of 5 minutes while being scanned (fmri) 5 - 30 min: fmri scan continues while subject lays still
  At t = 0, 2.5, 5, 10, 15 and 30 blood will be drawn and appetite ratings will be given.
  Interventions: Dietary Supplement: Chocolate milk - Oral Caloric
- Intra Gastric (Other): Subjects participated in a 35 min fmri scan. Intervention: intra-gastric infusion (naso-gastric tube) of 500 ml caloric load consisting of Nutricia Cholate Milk, over 5 min.
  While scanning:
  -5 - 0 min : baseline scan 0 - 5 min: intra-gastric infusion (naso-gastric tube) of 500 ml caloric load consisting of Nutricia Cholate Milk in a time frame of 5 minutes while being scanned (fmri) 5 - 30 min: fmri scan continues while subject lays still
  At t = 0, 2.5, 5, 10, 15 and 30 blood will be drawn and appetite ratings will be given.
  Interventions: Dietary Supplement: Chocolate milk - Intra Gastric Caloric

INTERVENTIONS:
Dietary Supplement: Water with guar gum - Non Caloric — Infusion 500 ml of water with 3 gram of guar gum through a naso-gastric tube directly into stomach during a fMRI scan.
  Other Names: Guar gum has the E number E412 and is allowed in the EU
  Arms: Control
Dietary Supplement: Chocolate milk - Oral Caloric — Ingestion of 500 ml of commercially available chocolate milk (Per 100mL; energy content of 354 kJ, 84 kcal, 3.5 g proteins, 12 g mono and disaccharide, 2.5 fat g, 0.5 g fibers) through a tube in the mouth during a fmri scan.
  Other Names: Chocomel®, FrieslandCampina, Ede, the Netherlands
  Arms: Oral ingestion
Dietary Supplement: Chocolate milk - Intra Gastric Caloric — Infusion of 500 ml of commercially available chocolate milk (Per 100mL; energy content of 354 kJ, 84 kcal, 3.5 g proteins, 12 g mono and disaccharide, 2.5 fat g, 0.5 g fibers) through a naso-gastric tube directly into stomach during a fMRI scan.
  Other Names: Chocomel®, FrieslandCampina, Ede, the Netherlands
  Arms: Intra Gastric

SUMMARY:
The amount and kind of food which is ingested influences the regulation of meal size. Neural signals from the gastrointestinal tract travel via the vagus nerve to the brainstem and thalamus, which projects to the rest of the brain, in particular the hypothalamus, amygdala and primary sensory cortices. In neuroimaging studies in which the stomach was distended with a gastric balloon activation was observed in the right insula, left posterior amygdala, left posterior insula, left inferior frontal gyrus and anterior cingulate cortex. So far, no study has examined the effects of the ingestion or infusion of a food on the brain. In addition to neural signals, hormonal signals are important for meal termination. Hormones like insulin, ghrelin and cholecystokinin interact with gastric as well as sensory signals in the process of satiation, which ultimately leads to meal termination. The aim of this study is to investigate the interaction between food administration, hormone responses and brain responses. To this end an oral or intra-gastric load will be administered while measuring brain activity (functional magnetic resonance imaging) and hormone concentrations. Subjects will participate in one trainings session and in three functional magnetic resonance imaging (fMRI) sessions (35-min fMRI scan). A training session will take 40-minutes and consists of placing a naso-gastric tube and ingesting 500 ml of chocolate milk orally. The fMRI sessions will consist of three conditions: in condition one (A) 500ml of chocolate milk will be administrated orally. In condition two (B) and three (C) an intra-gastric load of 500 ml is administrated.

DETAILED DESCRIPTION:
Study procedures

1. Screening: Before inclusion in the study, potential subjects will complete a screening questionnaire Subjects will then be informed about their eligibility. Also the procedure and risks will be explained. If they decide to participate, they will fill in and sign the standard MRI-screening form and the informed consent form. Also a training session date will be planed.
2. Training session: When subjects want to participate and match to the criteria a training session will be planned. During this training session a naso-gastric tube will be inserted by a qualified nurse (according to the "maagsonde-protocol" UMC Utrecht). After insertion of the tube subjects rest to allow water used to assist insertion of the tube to leave the stomach and to become comfortable with the tube. During this insertion the nurse and the subject can see if a subject can handle the naso-gastric tube and can or will participate in the study. Subjects will rate hunger, fullness, thirst, desire to eat, prospective consumption, nauseous, and anxiety on a VAS scale. To simulate the position in the MR scanner, subjects will be asked to lie down on a doctors table. A towel will be placed under need there right side, in this way the stomach will be more in the position when standing/sitting, this is to simulate normal gastric filling. A tube will be placed between the teeth of the subject (like a straw) after which an oral load of 500 ml will be ingested through the tube in the month. This ingestion will be driven by a pomp (100ml/min), which simulates a sip systematically. First 200 ml will be ingested, then there will be a pause of 30 seconds, second the next 150 ml will be pumped, following again a 30 second rest period, then the last 150 ml will be ingested. The subjects know the rate and speed of the sips and can stop the pomp on command when necessary. The subject will also hear a tone just before the sip is ingested. Here a subject learns to drink with a naso-gastric tube placed and when lying down. After ingestion the subjects will fill in the same questionnaire again. The naso-gastric tube will be removed after the rating. This training session will take about 40 minutes.
3. Assessments and procedures on the study days: All subjects will be asked to arrive in the morning after an overnight fast of at least 10 hours. The evening before the scan subjects will be ask to eat a standardized meal given by the researchers (AH kant & klaar). An appetite questionnaire will be filled in (hunger, fullness, thirst, desire to eat, quantity to eat, desire to eat something sweet or savory, nauseous, and anxiety). An intravenous cannula will be placed by a qualified person. Next, the naso-gastric tube will be placed (same procedure as training session). After the subject has been placed in the scanner (as in the training session with a towel under need there right side); one blood draw will be done for baseline measurements (e.g. glucose, insulin, cholecystokinin and ghrelin for every time point). The appetite questionnaire will be filled in again in the scanner. A reference and anatomic scan will be done. Now the fmri session begins; after five minutes of baseline scanning, food administration will start (t = 0). This consists of administration of the intra gastric load through the naso-gastric tube (caloric or non-caloric) or of ingestion of the caloric load through a tube (oral). Blood will be drawn at t = 2.5, t = 5, t = 10, t = 15 and at t = 30 min. Before every blood sample subjects will give fullness and nausea ratings. One of the researchers will stand next to the subject/scanner during the whole experiment. If aspiration occurs a researcher will be there to help immediately. The researchers also make sure a subject knows how to get out of the scanner as quick as possible if aspiration occurs. At t = 30 min the subject will be taken out the scanner and fill in the appetite questionnaire. The naso-gastric tube and intravenous cannula will be removed. Subsequently subjects will be provided with an ad libitum breakfast buffet at t = 45 min. Food weight and macro-nutrient intake will be recorded. After breakfast the appetite questionnaire is filled in once more.
4. Blood sampling and storage: On the study day, a 10 ml blood sample will be drawn by certified experienced medical personnel. Blood samples will be put on ice immediately and then centrifuged at 1730 × g for 10 min at 4 ˚C. Blood material from the collection tubes will be split into two portions and stored, one portion for the analyses and one portion as a backup. Blood serum will be stored at -80 ˚C at the Rudolf Magnus Institute until sample collection is complete. Only RMI laboratory personnel and the investigators will have access to the samples. Blood samples will be coded as follows: P01, P02, etc. The key to this code will only be known by the principal and medical investigators and not by the personnel performing the blood analyses. Samples will be kept for 10 years and then destroyed.
5. Naso-gastric tube: A qualified nurse will place the naso-gastric tube. The placement will go according to the 'maagsonde -protocol' (UMC Utrecht). After insertion of the tube subjects rest to allow water used to assist insertion of the tube to leave the stomach and to become comfortable with the tube.
6. Withdrawal of individual subjects: Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons. Each subject who does not complete the study for any reason will have a post-study screening by the end of the particular study day to ensure that the drop-out is not the result of a structural problem. Data of subjects who withdrew prematurely will be used for statistical analyses, as far as possible.
7. Replacement of individual subjects after withdrawal: In case subjects withdraw during the study (fMRI sessions), they will not be replaced. If a subject decides not to participate during the training session a new subject will be recruited.
8. Follow-up of subjects withdrawn from treatment: Subjects who withdraw from the study will not be followed up, unless they withdraw because of an adverse event.
9. Post-study screening: Subjects will be asked how they experienced the study procedures. This information, if the subject is willing to share it, will be used to evaluate (the burden of) the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (self-reported)
2. Males with age 18 and 35 year at day 01 of the study
3. Body Mass Index (BMI) between 20 and 25 kg/m2
4. Right-handed
5. Voluntary participation
6. Having given their written informed consent
7. Willing to comply with the study procedures
8. Willing to accept use of all anonymized data, including publication, and the confidential use and storage of all data
9. Willing to be informed about chance findings of pathology and approving of the disclosure of this information to the general physician (see Informed Consent)
10. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned (Belastingdienst)

Exclusion Criteria:

1. Smoking
2. Slimming or medically prescribed diet
3. Restrained eating
4. Having an eating disorder
5. Having a history of or current alcohol consumption > 28 units per week
6. Having a history of medical or surgical events that may significantly affect the study outcome, such as metabolic or endocrine disease, or any gastro-intestinal disorder
7. Use of medication, except aspirin/paracetamol
8. Claustrophobia
9. Having a taste or smell disorder or any neurological or psychiatric disorder
10. Having metal implants (i.e. pacemaker, metal joints, prostheses, etc.) or metal objects on the body which cannot be removed (i.e. piercing, hearing aid, brace, etc.)
11. Mental or physical status that is incompatible with the proper conduct of the study
12. Not having a general practitioner
13. Participation in any other clinical trial during this study.
14. Working at the Image Sciences Institute or the Radiology Department of the UMC Utrecht as employee or student.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline (when hungry) in brain activation during food infusion. | -5 tot 0 min and 0 to 5 min
  Brian activity is measured (fmri) non-stop. First 5 minutes refers to the baseline measurement (-5 - 0 min). Then food infusion starts (0 - 5 min). The differences in brain activation between the 5 min fmri measurement during baseline and food infusion is the main outcome.
Area under the curve of serum concentrations of hormones at a time frame of 30 minutes during and after food administration. | t = 0, 2.5, 5, 10, 15, and 30 minutes
  Change from baseline (t = 0; when hungry) in hormonal concentrations (glucose, insulin, cholecystokinin, ghrelin) during (0 - 5 min) and after (5 - 30 min) food administration. Measured at five time-points in 30 min.
Area under the curve in appetite ratings at a time frame of 30 min, as an effect of food administration. | t = 0, 2.5, 5, 10, 15 and 30 minutes
  Changes from baseline (t = 0; when hungry) in fullness, desire to eat and anxiety ratings during (0 - 5 min) and after (5 - 30 min) food administration. Measured at five time-points in 30 min.

SECONDARY OUTCOMES:
Energy intake (kJ) from the breakfast | at t = 45 min
  Amount of breakfast eaten after treatment
Changes from baseline in brain activity after food administration | 5 to 30 minutes
  After food administration brain activity was measured non-stop for 25 minutes. Activation in brain areas in this time frame were compared to baseline (when hungry).

CONTACTS AND LOCATIONS:
Overall Officials: Paul AM Smeets, Dr, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht - division Beeld, Utrecht, Netherlands

REFERENCES:
- [Derived] Spetter MS, de Graaf C, Mars M, Viergever MA, Smeets PA. The sum of its parts--effects of gastric distention, nutrient content and sensory stimulation on brain activation. PLoS One. 2014 Mar 10;9(3):e90872. doi: 10.1371/journal.pone.0090872. eCollection 2014. PMID 24614074